CLINICAL TRIAL: NCT06693531
Title: A U.S. Registry of Eosinophilic Esophagitis Patients Treated With DUPIXENT® As Standard of Care
Brief Title: A U.S. Registry of Eosinophilic Esophagitis Pediatric, Adolescent and Adult Patients Treated With DUPIXENT® As Standard of Care
Acronym: EDESIA
Status: Recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-EE-2328
Record Dates: First submitted 2024-10-30; First posted 2024-11-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EoE Patients treated with DUPIXENT®
  Interventions: Drug: dupilumab

INTERVENTIONS:
Drug: dupilumab — No investigational agents will be provided. Dupilumab will be prescribed as per usual clinical practice and will not be provided by the sponsor.
  Other Names: DUPIXENT®; REGN668; SAR231893

SUMMARY:
This observational research study is to better understand patients with eosinophilic esophagitis (EoE) who have recently been prescribed DUPIXENT® (dupilumab).

The purpose of this research study is to look at how DUPIXENT is used in normal care of patients with EoE.

Possible benefits to others include a better understanding of EoE and helping to inform research and clinical trial design leading to treatment decisions in this patient population going forward.

Patient questionnaires will measure the following:

* How EoE makes one feel
* EoE signs and/or symptoms, eg, how difficult it is to swallow
* How EoE affects quality-of-life
* How EoE impacts aspects of daily life
* How EoE symptoms have changed throughout the study

ELIGIBILITY:
Key Inclusion Criteria:

1. Initiating treatment with DUPIXENT® for EoE according to the USPI
2. Participants aged ≥12 years and caregivers or legal guardians of participants aged <12 years must be able to understand and complete registry-related questionnaires

Key Exclusion Criteria:

1. Patients who have a contraindication to DUPIXENT® according to the USPI
2. Treatment with DUPIXENT® within the 6 months prior to the screening assessment
3. Participation in an ongoing interventional study on or within 6 months of the baseline assessment. Once enrolled in registry, participation is allowed in other ongoing studies (at the discretion of the registry investigator)

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population comprises of patients (≥1 years old) who are initiating treatment with DUPIXENT® for EoE according to the United States Prescribing Information (USPI)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2030-05-22 (Estimated); Study Completion 2030-05-22 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristic of participants who receive dupilumab for EoE: Age | Baseline and up to 3 years after treatment initiation
Demographic characteristic of participants who receive dupilumab for EoE: Race | Baseline and up to 3 years after treatment initiation
Demographic characteristic of participants who receive dupilumab for EoE: Weight | Baseline and up to 3 years after treatment initiation
Demographic characteristic of participants who receive dupilumab for EoE: Height | Baseline and up to 3 years after treatment initiation
Disease characteristics of participants who receive dupilumab for EoE: Esophagogastroduodenoscopy (EGD) | Baseline and up to 3 years after treatment initiation
Disease characteristics of participants who receive dupilumab for EoE: Dilation/impaction history | Baseline and up to 3 years after treatment initiation
Disease characteristics of participants who receive dupilumab for EoE: Dietary interventions | Baseline and up to 3 years after treatment initiation
Disease characteristics of participants who receive dupilumab for EoE: Medical history | Baseline and up to 3 years after treatment initiation
EoE medication history of participant | Previous 1 year and up to 3 years after treatment initiation
Non-EoE medication history of participant | Previous 3 months and up to 3 years after treatment initiation
Prior dupilumab exposure history of participant | Baseline and up to 3 years after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (54):
- United States (54):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arizona Digestive Health/GI Alliance, Sun City, Arizona
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - University of California, San Francisco, Oakland, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - UConn Health - The Carole and Ray Neag Comprehensive Cancer Center, Farmington, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Orlando Health, Orlando, Florida
  - Emory Healthcare, Emory Clinic, Atlanta, Georgia
  - GI Care for Kids LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Comprehensive Gastrointestinal Health, LLC, Libertyville, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Kansas Gastroenterology LLC, Wichita, Kansas
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Boston Specialists, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - GI Associates and Endoscopy Center, Flowood, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Washington University in Saint Louis, St Louis, Missouri
  - Allergy Partners of N.J., P.C., Ocean City, New Jersey
  - Steven And Alexandra Cohen Children's Medical Center Of New York, Lake Success, New York
  - Weil Cornell Medicine NYP, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Gastroenterology Group of Rochester LLP, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Atrium Health / Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Susquehanna Research Group, Camp Hill, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Gastroenterology Clinical Research, Summerville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - GI Alliance, Southlake, Texas
  - Tanner Clinic, Layton, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Home Health Company, Seattle, Washington
  - Washington Gastroenterology, GIA, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin